CLINICAL TRIAL: NCT03403569
Title: Impact of Triptolide Wilfordii on Viral Suppression, Immune Recovery and Immune Activation Biomarkers in Treatment-naive HIV-1 Infection: a Randomized, Double-blinded, Placebo-controlled Study
Brief Title: Safety and Efficacy of Triptolide Wilfordii in New Onset HIV-1 Infection
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PekingUMCH record JS-985
Record Dates: First submitted 2018-01-11; First posted 2018-01-18 (Actual); Last update posted 2022-04-08 (Actual); Status verified 2020-03

CONDITIONS: HIV-infection/AIDS
Keywords: CD4 cell recovery; immune activation; anti-inflammation
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Triptolide Wilfordii Group (Experimental): 150 patients will be enrolled and be administrated with Triptolide Wilfordii 20mg three times a day(TID) per os combined with appropriate ART for 12 months.
  Interventions: Drug: Triptolide Wilfordii
- Placebo Oral Tablet Group (Placebo Comparator): 150 patients will be enrolled and be administrated with placebo per os combined with appropriate ART for 12 months.
  Interventions: Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: Triptolide Wilfordii — In addition to appropriate ART, Triptolide Wilfordii will be given to patients in the experimental group at a dosage of 20mg three times a day per os for 12 months.
  Arms: Triptolide Wilfordii Group
Drug: Placebo Oral Tablet — In addition to appropriate ART, placebo oral tablets will be given to patients in the experimental group at a dosage of 2 pills three times a day per os for 12 months.
  Arms: Placebo Oral Tablet Group

SUMMARY:
The traditional Chinese herbal medicine Triptolide Wilfordii has displayed remarkable effect on the treatment of autoimmune diseases such as rheumatoid arthritis. Now that immunosuppression therapy has recently become a new strategy for HIV infection, it's reasonable to expect the anti-inflammatory effect of Triptolide Wilfordii in HIV infected patients. So we designed a randomized, double-blinded, placebo-controlled study to explore the efficacy and safety of Triptolide Wilfordii in new-onset HIV infection.

DETAILED DESCRIPTION:
Acquired immune deficiency syndrome(AIDS) is a severe fatal disease caused by HIV infection. Despite viral suppression achieved, antiretroviral therapy(ART) cannot ameliorate HIV-induced immune activation and the consequent non-AIDS complications including cardiovascular, renal, hepatic diseases. Recently, immunosuppression therapy has become the focus since it can suppress exorbitant immune activation and inflammation so as to reduce the risk of non-AIDS cardiovascular and central neural system complications. Triptolide Wilfordii is a traditional Chinese herbal remedy and has long been used in the treatment of autoimmune diseases such as rheumatoid arthritis. Moreover, a recent study has shown that Triptolide Wilfordii combined with ART is associated with increased CD4 T cell counts and reduced immune activation in immunological non-responders, who were defined as patients with CD4 cell counts<350 cells/μl despite over 2 years of ART. Hence we expect Triptolide Wilfordii to bring up similar improvement in treatment naïve HIV infection. This randomized, double-blinded, placebo-controlled study is designed to investigate the safety and efficacy of Triptolide Wilfordii and hopefully provide evidence for a new treatment strategy.

ELIGIBILITY:
Inclusion Criteria:

* 18~65 years old;
* Male or female;
* Good adherence and promise to follow-up;
* Inform Consent signed;
* Positive for HIV antibody test or serum HIV-RNA positive for 2 times or more;

Exclusion Criteria:

* Present opportunity infection defined according to national AIDS treatment guideline or active opportunistic infection(not stable within 14 days ) within 3 months before recruitment or AIDS-related carcinoma;
* Hemoglobin (HGB) < 9 g/dl, white blood cell (WBC) < 3000/ul, granulin (GRN) < 1500 /ul, platelet (PLT) < 75000 /ul, Cr >1.5x upper limit of normal (ULN), ALT or AST or alkaline phosphatase (ALP) >3x ULN, total bilirubin (TBIL) >2x ULN;
* Pregnancy or breastfeeding;
* Woman with pregnancy plan;
* Severe organ dysfunction;
* Administration of immunosuppressor, immunomodulator(including thymocin) or systemic cytotoxic drugs within 6 months before recruitment.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 353 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
CD4 T cell counts and HIV RNA | Baseline, Week4, Week12, Week24, Week36, Week 48
  Compared to patients in placebo group, CD4 T cells of patients treated with Triptolide Wilfordii significantly increase and HIV RNA is reduced below 20 copies/ml.

SECONDARY OUTCOMES:
Immune activation | Baseline, Week4, Week12, Week24, Week36, Week 48
  Compared to patients in placebo group, immune activation index of patients treated with Triptolide Wilfordii decreases.
Inflammation level | Baseline, Week4, Week12, Week24, Week36, Week 48
  Compared to patients in placebo group, inflammation level of patients treated with Triptolide Wilfordii decreases.
HIV reservoir | Baseline, Week4, Week12, Week24, Week36, Week 48
  Compared to patients in placebo group, HIV reservoir of patients treated with Triptolide Wilfordii is reduced.

CONTACTS AND LOCATIONS:
Overall Officials: Wei Lyu, Principal Investigator — Department of Infectious Diseases, PekingUMCH
Locations (7):
- China (7):
  - Mengchao Hepatobiliary Hospital of Fujian Medical University, Fuzhou, Fujian
  - The Eighth People's Hospital of Guangzhou, Guangzhou, Guangdong
  - The Fourth Affiliated Hospital of Harbin Medical University, Harbin, Heilongjiang
  - The Sixth People's Hospital of Zhengzhou, Zhengzhou, Henan
  - Xixi Hospital of Hangzhou, Hangzhou, Zhejiang
  - Beijing YouAn Hospital, Capital Medical University, Beijing
  - Beijing Ditan Hospital, Capital Medical University, Beijing

IPD SHARING:
Plan to Share IPD: No